CLINICAL TRIAL: NCT00540319
Title: Prevention for Prenatal Health: the Health in Pregnancy (HIP) Study
Brief Title: The Health in Pregnancy (HIP) Study
Acronym: HIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA015597 (NIH); R01DA015597 (NIH)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy
Keywords: Risky behaviors; Prenatal care; Substance use; Domestic violence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: HIP — The Health in Pregnancy (HIP) computer program provides tailored, interactive "Video Doctor" counseling about behavioral risks, educational worksheets for the patients, and a cueing sheet for providers.

SUMMARY:
Pregnancy is a critical time to address preventable behavioral risks that pose serious threats to the health of both the mother and the developing fetus. We propose to conduct a randomized, controlled trial to determine the extent to which the Health in Pregnancy (HIP) program, a brief motivational intervention featuring a "Video Doctor," provider cueing sheets, and patient educational worksheets, can reduce pregnant women's cigarette smoking, alcohol drinking, illicit drug use, and domestic violence risks compared with usual care.

DETAILED DESCRIPTION:
Regular prenatal visits offer opportunities to deliver and reinforce risk reduction messages regarding tobacco, alcohol, or illicit drug use and domestic violence. Because health care providers may lack the time, comfort, or skills to screen or counsel their patients about these risks, innovative approaches are needed. Computer programs are increasingly used to assess risky behaviors and deliver individualized preventive interventions. We have designed a randomized, controlled trial to determine if a brief, interactive, multimedia intervention delivered on a laptop computer and integrated into routine prenatal care can reduce pregnant women's smoking, drinking, drug use, and experiences of domestic violence compared to usual care. To capitalize on health care providers' credibility, the multimedia intervention is delivered by an actor-portrayed "Video Doctor" programmed to respond to participant input, simulating a live interview. Pregnant women who receive prenatal care at one of the study sites and who consent to participate will be screened for substance use and domestic violence prior to a regularly scheduled medical appointment. Women who report one or more of these risks will be randomly assigned to the Intervention or Control group according to a blocked, stratified randomization plan. Participants in the Intervention group will receive the Health in Pregnancy (HIP) intervention, consisting of brief, multimedia counseling presented by a "Video Doctor" and an educational worksheet. Their provider will receive a "Cueing Sheet," which offers a brief summary of the patient's risk profile and suggests counseling statements. Components of the multimedia program will be tailored to each participant's risk profile and readiness to change. Women assigned to the Control group will complete a risk assessment than receive the usual care offered by the health care settings. Both Intervention and Control participants will complete two follow-up risk assessments at consecutive medical visits approximately four weeks apart. At the first follow-up session, Intervention participants will also receive "booster" risk reduction messages from teh video doctor. To determine the effect of the HIP program on patient-provider discussions, both Intervention and Control participants will complete a post-interview after their medical appointment. The post-interview will also assess the acceptability of the HIP program by participants. To determine the effect of teh program on participants' risky behaviors we will compare self-reported discussions, behavior change, and readiness to change at baseline and at a third session with the computer program. We expect that participants in the Intervention group will show significant reductions in risky behaviors compared to the Control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English speaking
* Pregnant and receiving prenatal care at a participating study site.

Exclusion Criteria:

* >25 weeks gestation at baseline session.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Elimination of cigarette smoking, alcohol drinking, and illicit drug use.
Reduction in frequency and/or severity of domestic violence.

SECONDARY OUTCOMES:
Patient-provider discussions of risks.
Measures of change in cigarette smoking, alcohol drinking, and illicit drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gerbert, PhD, Principal Investigator — University of California, San Francisco; Rebecca Jackson, MD, Study Director — San Francisco General Hospital
Locations (5):
- United States (5):
  - Highland Hospital, Oakland, California
  - San Francisco General Hospital, San Francisco, California
  - St. Luke's Hospital, San Francisco, California
  - UCSF Faculty Obstetrics and Gynecology Group, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3312043/